CLINICAL TRIAL: NCT07079709
Title: Returning to Work After Stress-Related Sick Leave: An Effectiveness Trial of Work-Focused Treatments in Primary Care
Acronym: ReWork
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Göteborg University (Other); Academic Primary Health Care Centre, SLSO, Region Stockholm (Unknown)
Responsible Party: Principal Investigator, Anna Finnes, PhD, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01713-01; 2023-01487 (Other Grant/Funding Number: Forte)
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Clinical Burnout; Exhaustion Disorder; Adjustment Disorder With Work Inhibition
Keywords: Work-focused CBT; WCBT; Sick leave; Clinical burnout; Cognitive behaviour therapy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled multi-center study, where control group centers providing treatment as usual are matched using the Care Need Index. Estimation of treatment effects will be conducted using either doubly robust inverse probability of treatment weights or targeted maximum likelihood estimation, depending on the outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WCBT (Experimental): Work-focused Cognitive Behaviour Therapy
  Interventions: Behavioral: Workfocused CBT
- Standard Care (Active Comparator): Standard Care is defined as care by the sick leave prescribing physician and the rehab coordinator. Other interventions such as psychological treatment, physiotherapy etc. may also be included in this arm.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: Workfocused CBT — In WCBT, the central idea is that CBT techniques can be applied in a work context with the aim of achieving both usual treatment goals related to symptoms and RTW. To ensure positive effects at both symptomatic and functional levels, a work perspective must be fully integrated into the intervention to optimize the treatment effect which demands collaboration with the sick leave prescribing doctor and the patient's employer. The protocol is based on principles of increasing return-to-work self-efficacy (RTW-SE). Work-specific components, such as work anamnesis, adjusting the difficulty of work tasks, and developing a return-to-work plan that includes recommendations for workplace accommodations, are integrated into all treatment sessions.
  Other Names: WCBT
  Arms: WCBT
Other: Standard Care (in control arm) — Standard Care is defined as care by the sick leave prescribing physician and the rehab coordinator. Other interventions such as psychological treatment, physiotherapy etc. may also be included in this arm.
  Arms: Standard Care

SUMMARY:
The goal of this clinical trial is to learn if work-focused cognitive behaviour (WCBT) works to treat patients on sick leave due to non-traumatic long-term stress-related disorders. The main questions it aims to answer are:

* Is WCBT more effective in improving work ability compared to standard care?
* Do participants in WCBT have less sick leave days than those in standard care?
* Is WCBT more effective in improving health outcomes and function than standard care?
* Is WCBT a more cost-effective treatment option than standard care? Researchers will compare WCBT to standad care to see if there are differences in effect.

Participants will participate in:

* WCBT
* Standard care

ELIGIBILITY:
Inclusion Criteria:

1. be on sick leave at least 50%
2. be diagnosed with a primary diagnosis adjustment disorder (F43.2-F.43.9) including exhaustion disorder (F43.8A)
3. be of working age (18-60 years)
4. be able to understand verbal and written Swedish or English
5. give informed consent

Exclusion Criteria:

1. other psychiatric conditions that require prioritization for immediate or simultaneous treatment: specifically, a current diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, or organic mental disorder; current high risk of suicide; or recent (within 3 months) history of substance use disorder)
2. other ongoing or recent (within 6 months) psychological treatment for stress-related disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
Work Ability Index (WAI) including Work Ability Score (WAS) | WAI: Baseline, 6 months, 1- and 2 year follow-up. WAS: every two weeks during the first six months.
  Self-reported change in work ability. WAI consists of 7 domains, 11 questions in total. WAS is the first question of WAI.

SECONDARY OUTCOMES:
Sick leave | The time horizon is two years prior to and five years after the date for inclusion in the study.
  Register data MiDAS from the Swedish Social Insurance Agency reflecting sickness absence - start- and stop date, both episodes and monthly panels for sickness benefit and activity compensation, diagnose, employment/occupation and paid out compensation.
Current work status and sick leave | Baseline, every two weeks until 6 months, 1- and 2-year follow-up.
  Participants will respond to the questions "Have you worked during the past week?" and "Are you currently on sick leave?". If yes, participants reports the proportion (25, 50, 75 or 100%) related to normal working hours.
Shirom-Melamed Burnout Questionnaire (SMBQ-6) | Baseline, every two weeks during 6 months, 1- and 2-year follow-up.
  Six items. Labels have been added to the original response scale. The participant can rate whether they experience the symptom "never", "almost never", "rarely", "sometimes" "fairy often", "almost always", "always".
Insomnia Severy Index (ISI) | Baseline, 6 months, 1- and 2 year follow-up.
  7 items.
Checklist Individual Strength | Baseline, 6 months, 1- and 2 year follow-up.
  This 20-item scale measures symptoms of fatigue. The participant is asked to rate statements and if he/she felt it during the last two weeks. Examples of questions are: "I feel tired", "I think I do a lot in a day", etc. The statements are rated on a 7-point scale with added labels as follows: "never true", "very rarely true", "rarely true", "sometimes true", "quite often true", "very often true", and "always true".
Patient Health Questionnaire (PHQ-9) | Baseline, 6 months, 1- and 2 year follow-up.
  Measures depressive symptoms. The occurrence of symptoms during the past two weeks is originally rated on a four-point scale labeled "not at all" to "nearly every day". To capture a more accurate estimation, an additional option category was added following a newly published study (see ref below). In addition, the highest option was adjusted from "nearly every day" to "every day" due to a high similarity between two options. The final response scale had the following five categories: "Not at all", "once or twice", "several days", "more than half the days", and "every day". The patient also rated how difficult those symptoms have made it for the participant to handle activities in everyday life.
  Ref: Makowski, D., Te, A., Neves, A., & Chen, S. A. (2024). Measuring Depression and Anxiety with 4 items? Adaptation of the PHQ-4 to increase its Sensitivity to Subclinical Variability. PsyArXiv. https://doi.org/10.31234/osf.io/436np
Generalized Anxiety Disorder Assessment (GAD-7) | Baseline, 6 months, 1- and 2 year follow-up.
  7 items. The occurrence of symptoms during the past two weeks is originally rated on a four-point scale labeled "not at all" to "nearly every day". To capture a more accurate estimation, an additional option category was added following a newly published study (see ref below). In addition, the highest option was adjusted from "nearly every day" to "every day" due to a high similarity between two options. The final response scale had the following five categories: "Not at all", "once or twice", "several days", "more than half the days", and "every day".
  Ref: Makowski, D., Te, A., Neves, A., & Chen, S. A. (2024). Measuring Depression and Anxiety with 4 items? Adaptation of the PHQ-4 to increase its Sensitivity to Subclinical Variability. PsyArXiv. https://doi.org/10.31234/osf.io/436np
Short Form Survey (SF-12) | Baseline, 6 months, 1- and 2 year follow-up.
  Measures quality of life in eight domains by 12 items.
Return to work Self-efficacy Scale | Baseline, 6 months, 1- and 2 year follow-up.
  Nine items from the original 11-item questionnaire were chosen, and items 3 and 11 were rewritten in order to achieve consistency in the wording. Item 2 was removed due to the overlap with item 4. Item 6 was removed since the question did not concern self-efficacy. Answers are rated on a 6-point labeled scale from "totally disagree" to "totally agree".
Work Phobia Questionnaire - short version | Baseline, every two weeks until 6 months, 1- and 2 year follow-up.
  Items 1, 2, 7, 9, 13 from the original questionnaire were chosen. In addition, labels were added to the six-point scale: "strongly disagree", "mostly disagree", "somewhat disagree", "somewhat agree", "mostly agree", "strongly agree".
Perceived Competence Scale | Baseline, 6 months, 1- and 2 year follow-up.
  4 items.
Psychological avoidance of stress - The psychological inflexibility in stress scale | Baseline, every two weeks during 6 months, 1- and 2 year follow-up.
  A subscale concering aviodance from the psychological inflexibility in pain scale was modified to measure aviodance related to stress. The word "pain" from the original scale was replaced by "stress". 8 items.
Lifestyle habits | Baseline, 6 months, 1- and 2 year follow-up.
  12 items.
Expactancy of improvement/Credibility | Only for the experimental group: 4 weeks after inclusion.
  The questions are inspired from the questionnaire "Credibility/Expectancy Questionnaire" but are designed for this study. 3 items: (I) how relevant the treatment seems at the moment, from "not at all" to "completely", (II) prediction of how the treatment will affect symptoms and (III) work ability, from "it will become much worse" to "it will be much better".
Working Alliance Inventory | Only for the experimental group: 4 weeks after baseline and 6 months post enrollment.
  6 items.
Client Satisfaction Questionnaire | Only for the intervention group: 6 months after enrollment.
  8 items.
Negative Effects Questionnaire - short version | 6 months post enrollment.
  Five questions are used from the original instrument, the Negative Effects Questionnaire. Included items: (I) the perception of being less competent, (II) worsening of the problem, (III) thoughts that the issue would not get better, (IV) feeling of shame due to having the treatment, (V) and development of dependency towards the therapist. If any of the statesmen were experienced, the participant rates how much it affects him/her on a scale from "not at all" to "extremely" and if it was caused by the treatment or other circumstances.

IPD SHARING:
Plan to Share IPD: Undecided